CLINICAL TRIAL: NCT02256306
Title: The PLasma for Alzheimer SymptoM Amelioration (PLASMA) Study: Intravenously-Administered Plasma From Young Donors for Treatment of Mild-To-Moderate Alzheimer's Disease
Brief Title: The PLasma for Alzheimer SymptoM Amelioration (PLASMA) Study
Acronym: PLASMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Alkahest, Inc. (Industry)
Responsible Party: Principal Investigator, Sharon Sha, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30350
Record Dates: First submitted 2014-09-25; First posted 2014-10-03 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Mild-To-Moderate Alzheimer's Disease; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Young Donor Plasma (Experimental): Subjects will receive 1 unit of plasma, once weekly for 4 weeks.
  Interventions: Other: Plasma

INTERVENTIONS:
Other: Plasma — 1 unit of Plasma From Young Donors (Male, aged 30 or younger)

SUMMARY:
The PLasma for Alzheimer SymptoM Amelioration (PLASMA) Study: Intravenously-Administered Plasma From Young Donors for Treatment of Mild-To-Moderate Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease (NIA-AA criteria)
* Mini-Mental State Examination (MMSE) score 12-24
* Availability of a study partner who knows the patient well and is willing to accompany the subject to all trial visits, to participate in questionnaires and to complete daily journal assessments

Exclusion Criteria:

* Pregnancy or unwilling to use adequate birth control method for duration of and 6 months beyond study participation
* Positive for Hepatitis B, Hepatitis C or HIV at screening
* Any other condition or situation that the investigator believes may interfere with the safety of the subject or the intent and conduct of the study
* Related to medical history:

  * Stroke
  * Anaphylaxis
  * Prior adverse reaction to any human blood product
  * Any history of a blood coagulation disorder or hypercoagulability
  * Congestive heart failure
  * Uncontrolled hypertension
  * Renal failure
  * Prior intolerance to intravenous fluids
  * Recent history of uncontrolled atrial fibrillation
  * IgA deficiency (by history)
* Related to medications or other treatments:

  * Any concurrent use of an anticoagulant therapy. Antiplatelet drugs (e.g., aspirin or clopidogrel) are acceptable
  * Initiation or change in the dosage of a cholinesterase inhibitor or memantine during the trial. A participant already on a cholinesterase inhibitor or memantine must be on a stable dose for at least one month prior to Screening
  * Concurrent participation in another treatment trial for Alzheimer's disease. If there was prior participation, the last dose of the investigational agent must have been at least 6 months prior to Screening
  * Treatment with any human blood product, including intravenous immunoglobulin, during the 6 months prior to Screening or during the trial
  * Concurrent daily treatment with benzodiazepines, typical or atypical antipsychotics, long-acting opioids, or other medications that, in the investigator's opinion, interfere with cognition. Intermittent treatment with short-acting benzodiazepines or atypical antipsychotics may be permitted, provided that no dose is administered within the 72 hours preceding any cognitive assessment
* Related to magnetic resonance imaging:

  * Claustrophobia
  * Any metallic surgical implant, like a pacemaker or clip that is incompatible with 3T MRI.

Certain metallic implants like joint replacements may be permitted, provided that specific manufacturer specifications are available and that the device is known to be safe for 3T MRI.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability, and number of subjects who comply with the research protocol as a measure of feasibility. | 9 weeks

SECONDARY OUTCOMES:
Change on the 13-item ADAS-Cog | 9 weeks
Change on the Trail-Making Test | 9 weeks
Change on the Clinical Dementia Rating scale Sum of Boxes (CDR-SB) | 9 weeks
Change on the Functional Activities Questionnaire (FAQ) | 9 weeks
Change on the Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) | 9 weeks
Change on the Geriatric Depression Scale | 9 weeks
Change on the Neuropsychiatric Inventory Questionnaire (NPI-Q) | 9 weeks

OTHER OUTCOMES:
Change in functional connectivity in the default mode network as assessed by resting state functional MRI | 9 weeks
Compositional assessment of plasma using in vitro analytical methods. The goal is to assess plasma components that might be associated with aging and/or Alzheimer's disease | 9 weeks
In vivo assessment of plasma samples to determine their potential histological effects on the hippocampus and their potential behavioral effects in animal models of cognition | 9 weeks
Differential effect of therapy on above outcomes as a function of ApoE genotype | 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] Sha SJ, Deutsch GK, Tian L, Richardson K, Coburn M, Gaudioso JL, Marcal T, Solomon E, Boumis A, Bet A, Mennes M, van Oort E, Beckmann CF, Braithwaite SP, Jackson S, Nikolich K, Stephens D, Kerchner GA, Wyss-Coray T. Safety, Tolerability, and Feasibility of Young Plasma Infusion in the Plasma for Alzheimer Symptom Amelioration Study: A Randomized Clinical Trial. JAMA Neurol. 2019 Jan 1;76(1):35-40. doi: 10.1001/jamaneurol.2018.3288. PMID 30383097